CLINICAL TRIAL: NCT06567353
Title: A Multi-mode Thermophysical Immunotherapy Study for Breast Cancer Liver Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0306v1.1
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Neoplasms; Liver Neoplasms; Metastasis
Keywords: Multi-mode Thermophysical Immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-mode ablation (Experimental): Subjects in this arm will receive image-guided multi-mode ablation.
  Interventions: Device: Multi-mode tumor treatment system
- Conventional radiofrequency ablation (Active Comparator): Subjects in this arm will receive image-guided radiofrequency ablation.
  Interventions: Device: Radiofrequency ablation therapeutic apparatus

INTERVENTIONS:
Device: Multi-mode tumor treatment system — All subjects are treated using the multi-mode tumor treatment system (Shanghai MAaGI Medical Technology Co., Ltd), with the treatment procedure conducted according to the temperature control mode for tumor ablation. The treatment procedure includes: rapid freezing of the tumor tissue to form an ice ball extending 5mm beyond the lesion, maintaining this state for 5 minutes, followed by thawing and rewarming; subsequently, RFA is performed to ensure complete ablation, with the ablation zone including a safety margin of 5-10mm around the tumor.
  Other Names: MTT-P1
  Arms: Multi-mode ablation
Device: Radiofrequency ablation therapeutic apparatus — All subjects are treated using the radiofrequency ablation therapeutic apparatus (MedSphere International (Shanghai) Co., Ltd.), with the treatment procedure conducted according to the preset power and time parameters to ensure a safety margin of 5-10mm.
  Other Names: S-1500
  Arms: Conventional radiofrequency ablation

SUMMARY:
This is a single-center, parallel-controlled clinical study designed to evaluate the safety, efficacy and impact on systemic anti-tumor immunity of a multi-mode integrated ablation system for the treatment of breast cancer liver metastases.

DETAILED DESCRIPTION:
This is a single-center, parallel-controlled clinical study. The study plans to enroll 10 subjects, with 5 in the multi-mode ablation group (experimental group) and 5 in the conventional radiofrequency ablation group (control group). The entire study includes a screening period, treatment period and follow-up period. By comparing multi-mode ablation with conventional radiofrequency ablation, the study aims to observe the efficacy, safety of the multi-mode ablation technique in subjects and its impact on the systemic anti-tumor immunity of subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, female gender;
2. Pathologically confirmed breast cancer liver metastases, in patients who are unable to tolerate or refuse surgical resection;
3. The number of lesions ≤ 3, with any single lesion diameter ≤ 4cm;
4. At least an interval of 1 month since the last local treatment;
5. Child-Pugh class A or B;
6. ECOG PS score ≤2, with an expected survival of >3 months.

Exclusion Criteria:

1. Liver function Child-Pugh class C;
2. Systemic widespread metastasis, with an expected survival of < 3 months;
3. History of esophageal (gastric fundus) variceal bleeding within the past month;
4. Dysfunction or failure of vital organs;
5. Presence of an active infection;
6. Irreparable coagulation abnormality;
7. Refractory massive ascites, pleural effusion or cachexia;
8. Pregnancy, altered consciousness or patients unable to cooperate with treatment;
9. Previously participated in other clinical studies and still within the follow-up period;
10. Any other factors deemed inappropriate for inclusion or that may affect the patient's participation in the study, as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Anti-tumor immune response | max 24 months
  The anti-tumor immune response refers to the effect and mechanism by which multi-mode ablation activates systemic persistent specific anti-tumor immunity, thereby inhibiting tumor metastasis and recurrence.

SECONDARY OUTCOMES:
6-Month Local Control Rate | 6 months
  6-month local control rate (LCR) refers to the proportion of patients in whom the primary tumor site lesions are completely suppressed after treatment among all treated patients six months after the start of treatment.
6-Month Progression-Free Survival | 6 months
  6-month progression-free survival (6-month PFS) refers to the percentage of patients who are alive without tumor progression or metastasis six months after the start of treatment.
1-Year Progression-Free Survival | 1 year
  1-year progression-free survival (1-year PFS) refers to the percentage of patients who are alive without tumor progression or metastasis one year after the start of treatment.
1-Year Overall Survival | 1 year
  1-year overall survival (1-year OS) refers to the percentage of patients who are still alive one year after the start of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China